CLINICAL TRIAL: NCT04655638
Title: High-Flow Nasal Therapy Versus Conventional Oxygen Therapy in Patients With COVID-19: A Randomized Controlled Trial (The COVID-HIGH Trial)
Brief Title: HFNT vs. COT in COVID-19
Acronym: COVID-HIGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Collaborators: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Responsible Party: Principal Investigator, Andrea Cortegiani, MD, Principal Investigator, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1th Dec 2020
Record Dates: First submitted 2020-12-03; First posted 2020-12-07 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Acute Respiratory Failure
Keywords: COVID-19; HFNT; Respiratory failure; COT; Oxygen; Pneumonia
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Pneumonia

STUDY DESIGN:
Intervention Model Description: Unblinded parallel-group randomized multicenter clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Therapy (Experimental): High flow nasal therapy
  Interventions: Device: High Flow Nasal Therapy
- Conventional Oxygen Therapy (Active Comparator): Conventional Oxygen therapy
  Interventions: Device: Conventional Oxygen Therapy

INTERVENTIONS:
Device: High Flow Nasal Therapy — High flow nasal therapy will be delivered by any device (standalone machine or ventilators able to deliver it). The initial flow rate will be set at 40 L/min and potentially increased up to 60 L/min, according to patient tolerance. Large-bore nasal prongs will be selected according to the size of patients' nostrils (i.e. 2/3 of the diameter of the patient's nostril). A surgical mask will be placed on top of the HFNT interface. The temperature will be set at 37°C or 34 °C according to the patient's comfort. The FiO2 will be adjusted to maintain SpO2 between 92-96%.
  Arms: High Flow Nasal Therapy
Device: Conventional Oxygen Therapy — Conventional Oxygen therapy will be delivered by any device or combination of devices used for delivering oxygen such as nasal cannula, Venturi Mask or Mask with or without a reservoir bag as per usual local practice. Oxygen flow will be titrated to achieve SpO2 between 92-96%.
  Arms: Conventional Oxygen Therapy

SUMMARY:
The aim of this unblinded parallel-group randomized multicenter clinical trial is to compare the clinical effectiveness of high flow nasal therapy (HFNT) with conventional oxygen therapy (COT) in patients with confirmed COVID-19 related acute hypoxemic respiratory failure.

DETAILED DESCRIPTION:
The interventions will be delivered in any hospital ward caring for COVID-19 patients.

The interventions under investigation will be high flow nasal therapy in comparison with conventional oxygen therapy.

HFNT will be delivered by any device (standalone machine or ventilators able to deliver it). The initial flow rate will be set at 40 L/min and potentially increased up to 60 L/min, according to patient tolerance. Large-bore nasal prongs will be selected according to the size of patients' nostrils (i.e. 2/3 of the diameter of the patient's nostril). A surgical mask will be placed on top of the HFNT interface. The temperature will be set at 37°C or 34 °C according to the patient's comfort. The FiO2 will be adjusted to maintain SpO2 between 92-96%. A feeding tube or a nasogastric tube will not represent a contraindication for the use of HFNT provided the patency of the used nostril.

Conventional Oxygen therapy will be delivered by any device or combination of devices used for delivering oxygen such as nasal cannula, Venturi Mask or Mask with or without a reservoir bag as per usual local practice. Oxygen flow will be titrated to achieve SpO2 between 92-96%.

Co-interventions: Patients potentially eligible for the study will be evaluated by the attending physicians and receive medical therapy based on the attending physician's decision and local protocols. Awake proning is allowed. Local protocols, including drugs and awake proning, will be discussed with the enrolling centers at the initiation visit, and adherence to WHO guidelines will be recommended. Written informed consent from all the patients will be collected.

Termination criteria & protocol violation: Criteria for weaning off COT or HFNT was at clinical discretion of the managing physician based on the improvement in oxygenation with ability to maintain SpO2 of 96% or greater with less than 0.30 of FiO2 or P/F > 300. The switch from COT to HFNT should be considered a protocol violation and should be based on clinical decision of the treating physician.

Criteria to be considered for escalation of treatment: 1) SpO2 ≤ 92% despite COT or HFNT or P/F ≤ 180 with FiO2 ≥ 50%, and 2) at least one of the following: respiratory rate ≥ 28 breaths/min, severe dyspnea, signs of increased work of breathing (e.g. use of accessory muscles). If the patient meets these criteria, escalation of treatment CPAP, NIV or IMV will be considered.

The choice of the type of escalating treatment will be a clinical decision of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Tested positive for SARS-CoV-2 using real-time reverse transcriptase PCR (RT-PCR) nasopharyngeal swabs
* Clinical signs of acute respiratory infection and radiological evidence of pneumonia
* Hospital admission in any ward or Emergency Department within 48 h
* SpO2 ≤ 92% or PaO2/FiO2 < 300 in room air and need for oxygen therapy according to clinical judgment, at the screening.

Exclusion Criteria:

* PaO2/FiO2 ≤ 200
* Respiratory rate ≥ 28 breaths/min and or severe dyspnea and or use of accessory muscles
* Need for immediate intubation or noninvasive ventilation (including CPAP) according to clinical judgment (e.g. clinical diagnosis of cardiogenic pulmonary edema, respiratory acidosis pH ≤ 7.3)
* Patients already on CPAP/NIV or HFNT at study screening
* Septic shock
* Evidence of multiorgan failure
* Glasgow Coma Scale < 13
* Inability to comprehend the study content and give informed consent
* PaCO2 > 45 mmHg, (if blood gas available) or history of chronic hypercapnia
* Patient already on long-term oxygen therapy (LTOT) or home NIV/CPAP (even if only overnight)
* Neuromuscular disease
* Limitation of care based on patients' or physicians' decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients needing escalation of treatment during hospital stay | 28 days
  Proportion of patients needing escalation of treatment (i.e. noninvasive ventilation - including CPAP - or intubation).

SECONDARY OUTCOMES:
Proportion of patients needing intubation during hospital stay | 28 days
Proportion of patients who receive CPAP during hospital stay | 28 days
  Proportion of patients who receive continuous positive airway pressure during hospital stay
Proportion of patients who receive NIV during hospital stay | 28 days
  Proportion of patients undergone noninvasive ventilation (e.g. BiLevel, PSV)
Proportion of patients admitted to intensive care unit during hospital stay | 28 days
Proportion of patients who terminate the study protocols for improvement | 28 days
Length of stay in hospital | 28 days
Time to escalation of treatment to CPAP/NIV during hospital stay | 28 days
Time to escalation of treatment to intubation/invasive ventilation during hospital stay | 28 days
Length of stay in ICU | 28 day
Days free from CPAP/NIV during hospital stay | 28 days
Ventilator-free days during hospital stay | 28 days
Oxygen-free days during hospital stay | 28 days
28-day mortality | 28 days from hospital admission
60-day mortality | 60 days from hospital admission
Hospital mortality | 28 days
Treatment interruption due to intolerance during study treatment | 28 days
Dyspnea score (BORG scale) during hospital stay | 28 days
  [0= no dyspnea to 10= severe dyspnea] - daily collection
National Early Warning Score 2 (NEWS2) during hospital stay | 28 days
  Daily collection of Six simple physiological parameters that form the basis of the scoring system: respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness or new confusion, temperature. A score is allocated to each parameter, with the magnitude of the score reflecting how extremely the parameter varies from the norm. The score is then aggregated and uplifted by 2 points for people requiring supplemental oxygen to maintain their recommended oxygen saturation. Range of values: 0 (best) - 23 (worst) points.
ROX index during hospital stay | 28 days
  SpO2/FiO2/Respiratory rate - daily collection

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cortegiani, MD, Principal Investigator — University of Palermo. Azienda Ospedaliera Policlinico Paolo Giaccone; Claudia Crimi, MD, Principal Investigator — Respiratory Medicine Unit, "Policlinico-Vittorio Emanuele San Marco" University Hospital
Locations (27):
- Greece (2):
  - Department of Anesthesiology, University of Thessaly, School of Health Sciences, Faculty of Medicine, Larissa
  - Department of Emergency Medicine, Faculty of Medicine, University of Thessaly, Larissa
- Italy (21):
  - UO di Pronto Soccorso e Medicina d'Urgenza Humanitas Research Hospital, Rozzano, Milano
  - U.O. di Medicina interna AULSS 7 Pedemontana, Bassano del Grappa, VI
  - Pulmonology and Respiratory Intensive Care Unit, S. Donato Hospital, Arezzo, Italy, Arezzo
  - Institute of Respiratory Disease, Department of Basic Medical Science, Neuroscience and Sense Organs, University of Bari, Bari
  - Ospedale di Carpi, Carpi
  - Respiratory Medicine Unit, "Policlinico-Vittorio Emanuele San Marco" University Hospital, Catania, Italy, Catania
  - UO di Medicina d'Urgenza AOU Policlinico Vittorio Emanuele San Marco di Catania, Catania
  - Respiratory Section, Department of Translational Medicine, University of Ferrara. AOU Ferrara Arcispedale S. Anna. U.O. Pneumologia, Ferrara
  - Department of Medical and Surgical Sciences, University of Foggia. Institute of Respiratory Diseases, University Hospital 'Policlinico Riuniti', Foggia
  - UO di Pneumologia ASST Fatebenefratelli Sacco, Milan
  - AO DEI COLLI - PO Monaldi UO di Pneumologia e Fisiopatologia Respiratoria, Napoli
  - AOU San Luigi Gonzaga, Orbassano
  - Emergency Department, "S. Maria della Misericordia" Hospital, Perugia, Italy., Perugia
  - U.O. di Pneumologia Azienda USL di Pescara, Pescara
  - UO di Pronto Soccorso e Medicina d'Urgenza AUSL Romagna PO Rimini Ospedale "Inferni", Rimini
  - U.O. di PneumoCovid Azienda Ospedaliera San Giovanni di Roma, Roma
  - UO di Pneumologia Ospedale S. Bartolomeo, Sarzana
  - Department of Pneumology, A.O.U. Città della Salute e della Scienza of Turin, Italy., Turin
  - U.O. di Pneumologia ASST Settelaghi Ospedale Circolo Fondazione Macchi, Varese
  - U.O. Medicina Respiratoria del Policlinico G.B. Rossi, Verona
  - U.O. di Pneumotisiologia Ospedale di Vittorio Veneto Azienda ULSS 2 Marca Trevigiana, Vittorio Veneto
- Department of Pneumonology, Faculty of Medical Sciences in Katowice, Medical University of Silesia, Katowice, Poland
- Hospital Prof. Doutor Fernando Fonseca, Pneumologia, Amadora, Portugal
- Hospital Parc Taulí de Sabadell, Pneumologia, Sabadell, Spain
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Rochwerg B, Einav S, Chaudhuri D, Mancebo J, Mauri T, Helviz Y, Goligher EC, Jaber S, Ricard JD, Rittayamai N, Roca O, Antonelli M, Maggiore SM, Demoule A, Hodgson CL, Mercat A, Wilcox ME, Granton D, Wang D, Azoulay E, Ouanes-Besbes L, Cinnella G, Rauseo M, Carvalho C, Dessap-Mekontso A, Fraser J, Frat JP, Gomersall C, Grasselli G, Hernandez G, Jog S, Pesenti A, Riviello ED, Slutsky AS, Stapleton RD, Talmor D, Thille AW, Brochard L, Burns KEA. The role for high flow nasal cannula as a respiratory support strategy in adults: a clinical practice guideline. Intensive Care Med. 2020 Dec;46(12):2226-2237. doi: 10.1007/s00134-020-06312-y. Epub 2020 Nov 17. PMID 33201321
- [Background] Crimi C, Noto A, Cortegiani A, Impellizzeri P, Elliott M, Ambrosino N, Gregoretti C. Noninvasive respiratory support in acute hypoxemic respiratory failure associated with COVID-19 and other viral infections. Minerva Anestesiol. 2020 Nov;86(11):1190-1204. doi: 10.23736/S0375-9393.20.14785-0. Epub 2020 Aug 5. PMID 32756535
- [Background] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: Guidelines on the Management of Critically Ill Adults with Coronavirus Disease 2019 (COVID-19). Crit Care Med. 2020 Jun;48(6):e440-e469. doi: 10.1097/CCM.0000000000004363. PMID 32224769
- [Background] Braunlich J, Mauersberger F, Wirtz H. Effectiveness of nasal highflow in hypercapnic COPD patients is flow and leakage dependent. BMC Pulm Med. 2018 Jan 24;18(1):14. doi: 10.1186/s12890-018-0576-x. PMID 29368599
- [Derived] Crimi C, Noto A, Madotto F, Ippolito M, Nolasco S, Campisi R, De Vuono S, Fiorentino G, Pantazopoulos I, Chalkias A, Libra A, Mattei A, Scala R, Clini EM, Ergan B, Lujan M, Winck JC, Giarratano A, Carlucci A, Gregoretti C, Groff P, Cortegiani A; COVID-HIGH Investigators. High-flow nasal oxygen versus conventional oxygen therapy in patients with COVID-19 pneumonia and mild hypoxaemia: a randomised controlled trial. Thorax. 2023 Apr;78(4):354-361. doi: 10.1136/thoraxjnl-2022-218806. Epub 2022 May 17. PMID 35580898